CLINICAL TRIAL: NCT01931683
Title: Effect-site Concentration of Remifentanil for Smooth Removal of the LMA From Propofol Anesthesia
Brief Title: Dosing Study of Remifentanil for Smooth Removal of the Laryngeal Mask Airway (LMA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Associate professor, Ajou University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AJIRB-MED-CT4-13
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Drug Usage
Keywords: LMA removal; remifentanil; propofol
MeSH Terms: interventions — Remifentanil; Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- remifentanil (Experimental): LMA removal was accomplished when remifentanil was maintained a predetermined concentration throughout the emergence periods.
  Interventions: Drug: remifentanil; Device: laryngeal mask airway (LMA)

INTERVENTIONS:
Drug: remifentanil — The concentration of remifentanil was determined by modified Dixon's up-and-down method, starting from 1.0 ng/ml (0.2 ng/ml as a step size)
  Other Names: Ultiva
Device: laryngeal mask airway (LMA) — LMA was removed when the patients opened their eyes, and spontaneous respiration and adequate tidal volume and ventilatory frequency were confirmed

SUMMARY:
The investigators attempted to determine the optimal effect-site concentration of remifentanil for smooth removal of the LMA from propofol anesthesia.

DETAILED DESCRIPTION:
At the end of the surgery, propofol infusion was stopped and remifentanil was titrated to predetermined (initial concentration 1.0 ng/ml for the first patient). LMA removal was performed when the patients opened their eyes and spontaneous respiration and adequate tidal volume and ventilatory frequency were confirmed.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-II patients undergoing general anesthesia for short elective surgery (<1 hr)

Exclusion Criteria:

* G-E reflux
* obesity (BMI>30)
* anticipated difficult airway

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2013-10; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
smooth removal of LMA | from end of surgery to removal of LMA (participants will be followed for the emergence periods, an expected average of 15 min).
  the response of patients to the removal of LMA (classified as either 'success [smooth emergence]' or 'failure') during infusion of remifentanil.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Yeop Kim, MD, Study Director — Ajou University School of Medicine
Locations (1):
- Ajou University School of Medicine, Suwon, South Korea